CLINICAL TRIAL: NCT05678114
Title: The Effect of Inositol Treatment in Women With PCOS of Different Phenotype
Brief Title: Inositol Treatment in Different Type of PCOS Phenotype
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lo.Li.Pharma s.r.l (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ins-PCOSphenotype
Record Dates: First submitted 2022-12-21; First posted 2023-01-10 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Inositol

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hyperandrogenic PCOS (Experimental)
  Interventions: Dietary Supplement: Myo-inositol
- Non-hyperandrogenic PCOS (Experimental)
  Interventions: Dietary Supplement: Myo-inositol

INTERVENTIONS:
Dietary Supplement: Myo-inositol — Myo-inositol (4g/die)

SUMMARY:
Evaluation of the efficacy of inositol treatment in women with PCOS in relation to the phenotype (according to the Rotterdam Criteria)

ELIGIBILITY:
Inclusion Criteria:

* women with PCOS of any phenotype

Exclusion Criteria:

* hormonal treatment (such as contraceptive pill)
* use of supplements containing myo-inositol
* severe co-morbidities

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — women with polycystic ovary syndrome
Enrollment: 120 (Actual)
Dates: Start 2022-12-21 (Actual); Primary Completion 2023-04-28 (Actual); Study Completion 2023-05-12 (Actual)

PRIMARY OUTCOMES:
Regularization of the menstrual cycle | Change from baseline number of women with irregular menstrual cycle at 4 months
  Number of women with regular/altered menstrual cycle

CONTACTS AND LOCATIONS:
Locations (1):
- Clinica Alma Res, Roma, Italy

IPD SHARING:
Plan to Share IPD: No